CLINICAL TRIAL: NCT06197100
Title: Effectiveness of Supportive Care Training Given to Mothers of Babies With Infant Colic: Randomized Controlled Study
Brief Title: Supportive Care Training Given to Mothers of Babies With Infants Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Elif Tuba KOC, Child Health and Diseases Nursing Department President, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AhiEvranU-UTubaKOÇ-002
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Mothers; Infantile Colic
Keywords: infant; Infantile Colic; support intervention; mothers; Breast Feeding; crying baby
MeSH Terms: conditions — Colic; Breast Feeding

STUDY DESIGN:
Intervention Model Description: there are three sections to it, and they will all be finished simultaneously. This is not a study of drugs or devices. The two arms of the study are Supportive care training, and control groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supportive care training (Experimental): Training in supportive care will be given to the experimental group (Training group). The mothers will also receive a training booklet from the researchers. The training booklet covers burping newborns, massage, and nourishment for mothers. In addition, mothers will be observed nursing their children, and appropriate breastfeeding instruction will be given if the baby's holding position is a problem. Over the course of a week, the supportive care training intervention will be given in three modules to the experimental group. The interventions will be carried out by the first investigator, a pediatric nursing specialist.
  Interventions: Other: Supportive care training
- control groups (Active Comparator): An educational pamphlet regarding mother-baby nutrition and how to soothe a crying infant will be distributed to mothers in the control group.
  Interventions: Other: control grups

INTERVENTIONS:
Other: Supportive care training — The program includes breastfeeding teaching, baby massage, managing gas issues (shaking, white noise), and nutrition for mothers.
  Other Names: The researcher will conduct training with the supporting training group and provide them with a booklet that they have created.
  Arms: supportive care training
Other: control grups — Mothers in this group will be given an educational brochure containing information about colic.
  Other Names: educational brochure
  Arms: control groups

SUMMARY:
Infantile Colic is a non-pathological condition that causes babies to cry excessively throughout their first few months of life. It has a prevalence of 15-30% and is defined by excessive sobbing for at least 3 hours per day, 3 days per week for around 3 weeks.

Excessive sobbing, blushing, parachroma around the lips, bloating in the abdomen, drawing the legs into the abdomen, coldness at the ends, and fisting of the hands are all symptoms of infantile colic. Another significant clinical aspect of Infantile Colic is its protracted, difficult to soothe, and inexplicable nature. Infantile Colic is thought to have a cicadian pain cycle that begins in the evening.

Infantile Colic is a non-pathological condition that causes babies to cry excessively throughout their first few months of life. It has a prevalence of 15-30% and is defined by excessive sobbing for at least 3 hours per day, 3 days per week for around 3 weeks.

Excessive sobbing, blushing, parachroma around the lips, bloating in the abdomen, drawing the legs into the abdomen, coldness at the ends, and fisting of the hands are all symptoms of infantile colic. Another significant clinical aspect of Infantile Colic is its protracted, difficult to soothe, and inexplicable nature. Infantile Colic is thought to have a cicadian pain cycle that begins in the evening.

Anxiety and stress that arise during the postpartum period cause a variety of issues in both the mother and the baby, and have a negative impact on the mother-baby bond as well as the mother's care and parenting skills. Sleep deprivation, sleep disturbance, and exhaustion are said to be caused by the sensation of not being able to meet the child's demands. It has been found that as parental stress levels rise, the gut flora deteriorates, and increasing cortisol in breast milk increases the baby's crying attacks. Colic and excessive crying are also risk factors for unfavorable parent-infant interactions. Infantile Colic has been shown to have a negative impact on children's health in the short and long term for all of these reasons. As a result, healthcare experts must devise therapies to lessen the painful impact of Infantile Colic on babies and their families. As a result, the purpose of this study was to see how supportive care training for parents affected the colic levels of babies with Infantile Colic, as well as mothers' perceptions of nursing and parental self-efficacy.

DETAILED DESCRIPTION:
Research hypotheses; Supportive care training for mothers of babies with infantile colic H1: Has an effect on the average nursing self-efficacy scores of moms of newborns with infantile colic.

H2: It affects the parental self-efficacy score averages of moms of infantile colic kids, H3: It influences the colic scores of infantile colic babies.

MATERIALS AND METHODS Type of Research Research; It was planned as a pretest-posttest randomized controlled experimental study.

Purpose of the research Research; It was planned to determine the effect of the educational supportive care program for parents on the colic levels of babies with Infantile Colic, the parenting self-efficacy of mothers and the level of mother-infant attachment.

Place and Characteristics of the Research It will be held at the Pediatrics Polyclinic of Kırşehir Ahi Evran University Training and Research Hospital. There are 6 specialist physicians working in the pediatric outpatient clinic.

At the hospital where the research will be conducted, the pediatrician performs a detailed history and physical examination to diagnose infantile colic and identify symptomatic findings. It questions when the crying spells start during the day, tracking the duration of crying, and the baby's behavior. During a complete physical examination, the baby's weight gain, nutrition, defecation pattern, fever and illness are questioned and monitored. Factors that may affect the baby's infantile colic status, such as the baby's diarrhea, eczema, cow's milk protein allergy, lactose intolerance, and mother's smoking, are questioned. In addition, other problems and diseases in the baby's intestines are also questioned. After the history and physical examination are completed by the pediatrician, the baby is diagnosed with infantile colic according to the Rome IV diagnostic criteria.

Design and Blinding This prospective, randomized controlled study is planned to be carried out at Kırşehir Ahi Evran University Training and Research Hospital Pediatrics outpatient clinic between March 2024- August 2024. The study will be conducted based on the CONSORT protocol.

The study population will consist of 1-3 month old babies and their mothers who applied to the Pediatrics outpatient clinic with complaints of restlessness and crying between marc March 2024- August 2024 and were diagnosed with Infantile Colic by the physician, and who meet the research criteria and are selected by randomization. Similar studies were taken into account for the sample of the study. Then, a power analysis will be performed by a statistician using the G*Power program. Thus, the number of samples to be taken into the experimental and control groups will be determined.

Babies and mothers who meet the inclusion criteria will be randomly assigned to experimental and control groups through the online program (http://www.randomizer.org).

Blinding in the study included the parents of the babies included in the study, a pediatrician from the researchers, and a specialist nurse. The first researcher, who only implements the supportive education program, is not blind, so the pre-test post-test evaluation of the study will be collected independently by the second researcher, a specialist nurse. Additionally, the evaluation will be analyzed by an independent statistician. Therefore, the current study will be conducted as a double-blind randomized controlled trial.

Research Inclusion Criteria

* Gestational week >37, birth weight >2500g,
* No congenital anomalies related to the digestive system or nutrition,
* Postnatal age of 1-3 months,
* Not receiving colic treatment,
* Diagnosed with Infantile colic by a pediatrician,
* Babies who are exclusively breastfed,
* Mothers of these babies who are over 18 years old, do not use sedative or antiepileptic drugs, can understand and communicate in Turkish, have no mental disabilities, and volunteer to participate in the study will be included in the research.

Research Exclusion Criteria Babies whose gestational week is ≤ 37 and birth weight ≤ 2500g, who have metabolic diseases and congenital anomalies of the digestive system, who are being treated for colic, who are not breastfed, whose postnatal age is less than 1 month and more than 3 months, and who are under 18 years of age, who do not take antibiotics, sedatives or Mothers who use an antiepileptic type of medication, have communication problems and mental disabilities, and who do not consent to the research will not be included in the study.

Experimental Control Group Matching Criteria of the Research In randomized controlled studies, the number of participants in the groups is expected to be equal or balanced, as well as to be similar in terms of prognostic factors. Therefore, mothers in the experimental and control groups; Babies will be selected similar in terms of age, gender, educational status, marital status and number criteria, and babies will be selected in terms of birth week and birth weight. Stratified randomization will be performed in the study according to these criteria.

Data Collection Tools Data of the research; It will be collected by face-to-face interview with the parent, using the Child and Parent Introduction Form, Breastfeeding Self-Efficacy Scale and Perceived Maternal Parenting Self-Efficacy Scale.

Child and Parent Identification Form This form consists of 4 questions regarding the mother's age, education level, medications used and the baby's birth date.

Breastfeeding Self-Efficacy Scale It is a scale consisting of 33 items developed by Dennis (1999). It consists of two sub-dimensions to determine mothers' breastfeeding skills, beliefs and behaviors regarding breastfeeding. The validity and reliability study of the Turkish form of the scale was conducted by Ekşioğlu and Çeber .

* Technical sub-dimension: It is aimed at determining the mother's breastfeeding skills, such as being able to place the baby on the breast, giving appropriate positioning, recognizing the signs of good breastfeeding, and weaning the baby from the breast.
* Sub-dimension related to personal thoughts: It consists of items including the mother's willingness to feed her baby with breast milk, her belief that she will have milk, not using formula or bottle, and her beliefs and behaviors regarding coping with breastfeeding difficulties.

The scale prepared as a five-point Likert type; I never trust myself, I don't trust myself very much, I sometimes trust myself, I trust myself most of the time, I always trust myself. As the total score on the scale increases, breastfeeding self-efficacy also increases. The lowest score is 33 and the highest score is 165.

Perceived Mother Parenting Self-Efficacy Scale It was developed by Barnes and Adamson-Macedo in 2007 to determine the self-efficacy levels of women who gave birth prematurely. The scale is designed as a four-category scale type; It is an 18-item scale consisting of positive items such as "strongly disagree = 1, disagree = 2, agree = 3, strongly agree = 4". The validity and reliability study of the scale in Turkey was conducted by Verici and Kavlak in 2021. The Cronbach alpha coefficient examined for the internal consistency reliability of the scale was found to be 0.943. A minimum of 18 points and a maximum of 72 points are obtained from the Perceived Mother Parenting Self-Efficacy Scale. An increase in the score obtained indicates that the mother's self-efficacy level increases.

Infant Colic Scale (Appendix-4) The Infant Colic Scale was developed in 2002 by Marsha L. Cirgin Ellet and her colleagues to assist healthcare professionals in diagnosing and evaluating colic. The scale consists of 5 sub-dimensions and 22 questions: Cow's milk/soy protein allergy/intolerance, immature digestive system, immature central nervous system, difficult baby, parent-infant interaction + problematic baby. The Cronbach alpha coefficient of the scale was found to be 0.73.

The validity and reliability study of the scale in Turkey was conducted by Çetinkaya and Başbakkal in 2006. The Cronbach alpha coefficient examined for the internal consistency reliability of the scale was found to be 0.73 (16). The items of the infant colic scale were evaluated on a 6-point Likert scale. Scale items were rated with Likert-type scoring ranging from 1 to 6. The rating was made from 1 (strongly disagree) to 6 (strongly agree). Negative questions were reverse coded for consistency in interpretation of scores. Item 3 in the immature digestive system sub-dimension, items 7, 8, 9 in the immature central nervous system sub-dimension, items 13, 14, 15 in the difficult baby sub-dimension, item in the parent-infant interaction+problem baby sub-dimension. Items 17 and 19 were reverse coded. A low mean score from the scale indicates that colic has decreased, while a high mean score indicates that colic has increased.

Pre-Application A preliminary application will be made with a total of 10 mothers who are not included in the study sample, and the clarity and functionality of the data collection tools will be evaluated. After the preliminary application, necessary corrections will be made to the data collection tools.

APPLICATION Study data will be collected between February 2022 and June 2023. The study group (training group or control group) to which the mothers of infants with infantile colic will be included will be determined by computer using a simple random sampling method. The pre-test of the study will be administered to the experimental and control groups with the Child and Parent Introductory Form, Breastfeeding Self-Efficacy Scale and Perceived Mother Parenting Self-Efficacy Scale before the intervention, and the post-test will be administered immediately and 1 week after the intervention ends.

Supportive care training will be given to the experimental group (Training group). In addition, the booklet prepared by the researchers for the training will be given to the mothers. The supportive care training intervention to be applied to the experimental group is planned to be implemented in 3 modules for 1 week. Interventions will be carried out by the first investigator, a specialist pediatric nurse. Information regarding supportive care training is included in the appendix.

Mothers in the control group will be given an educational brochure containing information on mother-baby nutrition and comforting the baby when crying.

ELIGIBILITY:
Inclusion Criteria:

* Gestational week >37, birth weight >2500g,
* No congenital anomalies related to the digestive system or nutrition,
* Postnatal age of 1-3 months,
* Not receiving colic treatment,
* Diagnosed with Infantile colic by a pediatrician,
* Babies who are exclusively breastfed,
* Mothers of these babies who are over 18 years old, do not use sedative or antiepileptic drugs, can understand and communicate in Turkish, have no mental disabilities, and volunteer to participate in the study will be included in the research.

Exclusion Criteria:

* Gestational week ≤ 37 and birth weight ≤ 2500g,
* Those with metabolic disease and congenital anomalies of the digestive system,
* treated for colic,
* not breastfed,
* Babies whose postnatal age is less than 1 month and more than 3 months

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-efficacy | before intervention/15 days after the intervention
  Breastfeeding Self-efficacy Scale: It is a scale consisting of 33 items developed by Dennis (1999). It consists of two sub-dimensions to determine mothers' breastfeeding skills, beliefs and behaviors regarding breastfeeding.
Perceived Maternal Parenting Self-Efficacy | before intervention/15 days after the intervention
  Perceived Maternal Parenting Self-Efficacy Scale: It was created in 2007 by Barnes and Adamson-Macedo to assess the degree of self-efficacy among women who had babies early. The scale yields a minimum of 18 points and a maximum of 72 points. A rise in the score signifies an increase in the mother's degree of self-efficacy.
Infant Colic | before intervention/15 days after the intervention
  The Infant Colic Scale was developed in 2002 by Marsha L. Cirgin Ellet and her colleagues to assist healthcare professionals in diagnosing and evaluating colic. The scale consists of 5 sub-dimensions and 22 questions: Cow's milk/soy protein allergy/intolerance, immature digestive system, immature central nervous system, difficult baby, parent-infant interaction + problem baby.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Despriee AW, Magi CO, Smastuen MC, Glavin K, Nordhagen L, Jonassen CM, Rehbinder EM, Nordlund B, Soderhall C, Carlsen KL, Skjerven HO. Prevalence and perinatal risk factors of parent-reported colic, abdominal pain and other pain or discomforts in infants until 3 months of age - A prospective cohort study in PreventADALL. J Clin Nurs. 2022 Oct;31(19-20):2784-2796. doi: 10.1111/jocn.16097. Epub 2021 Oct 26. PMID 34704296
- [Background] Hjern A, Lindblom K, Reuter A, Silfverdal SA. A systematic review of prevention and treatment of infantile colic. Acta Paediatr. 2020 Sep;109(9):1733-1744. doi: 10.1111/apa.15247. Epub 2020 Jun 2. PMID 32150292
- [Background] Shirazinia R, Golabchifar AA, Fazeli MR. Efficacy of probiotics for managing infantile colic due to their anti-inflammatory properties: a meta-analysis and systematic review. Clin Exp Pediatr. 2021 Dec;64(12):642-651. doi: 10.3345/cep.2020.01676. Epub 2021 Apr 12. PMID 33848417
- [Background] Zeevenhooven J, Browne PD, L'Hoir MP, de Weerth C, Benninga MA. Infant colic: mechanisms and management. Nat Rev Gastroenterol Hepatol. 2018 Aug;15(8):479-496. doi: 10.1038/s41575-018-0008-7. PMID 29760502
- [Background] Khajeh M, Sadeghi T, Ramezani M, Derafshi R. Effect of mothers' educational supportive care program on pain intensity and crying duration caused by colic pain in infants aged 1-5 months. Evid Based Care J. 2019;9(1):7-15.
- [Background] Hechler C, Beijers R, Riksen-Walraven JM, de Weerth C. Are cortisol concentrations in human breast milk associated with infant crying? Dev Psychobiol. 2018 Sep;60(6):639-650. doi: 10.1002/dev.21761. Epub 2018 Jul 1. PMID 29961271
- [Background] Ong TG, Gordon M, Banks SS, Thomas MR, Akobeng AK. Probiotics to prevent infantile colic. Cochrane Database Syst Rev. 2019 Mar 13;3(3):CD012473. doi: 10.1002/14651858.CD012473.pub2. PMID 30865287
- [Background] Hatch M, Landy K. Do parent training programs reduce crying time in infants with and without colic? Evidence-Based Pract. 2022;25(6):16-7.